CLINICAL TRIAL: NCT03748992
Title: A Proof of Concept Study of Inhaled Nitric Oxide for Adults With Pulmonary Non-Tuberculous Mycobacterial Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro 00081838
Record Dates: First submitted 2018-11-19; First posted 2018-11-21 (Actual); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Nontuberculous Mycobacterium Infection
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- gNO (Experimental): Subjects will be receiving nitric oxide every week day for 3 weeks.
  Interventions: Drug: gNO

INTERVENTIONS:
Drug: gNO — This is a proof-of-concept study in which all subjects will be treated with gNO (i.e. no control) to see if there can be a microbiological effect by conversion to negative sputum cultures and how long that effect can be sustained following treatment.
  Participants will be treated for 3 weeks (5 days per week), Monday through Friday, and followed monthly for 3 months.
  The treatment period includes a physical exam, vital signs, blood tests, echocardiogram, spirometry test, sputum sample, questionnaires, and the inhalation gas treatment. During the inhalation gas treatment, participants will wear a face mask (similar to an oxygen mask) and will be given nitric oxide gas through the participants nose for three treatments with fifty minutes each time. They will then be followed up monthly during the Follow-up period with tests that include a physical exam and questionnaires.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of open-label exposure of gNO in patients with NTM lung disease. Subjects will receive the study drug by inhaling through a nasal mask. Subjects will be treated for 3 weeks (5 days per week) and followed monthly for 3 months.

ELIGIBILITY:
Inclusion Criteria:

Subjects are >18 years of age and able to provide informed consent.

Subjects have NTM lung disease as defined by each of the following:

Sputum cultures positive for NTM (MAC or M abscessus) Radiologic studies that demonstrate features consistent with disease such as nodular bronchiectasis and/or cavities Symptoms consistent with disease including respiratory (e.g. cough, sputum production, hemoptysis, chest pain) and constitutional (e.g. fevers, night sweats, fatigue, myalgias, arthralgias, weight loss) Subjects are able to produce sputum for culture (either spontaneous or induced).

Subjects have a history of persistently positive sputum cultures for NTM defined as >4 number of cultures over 24 months with >75% positive AND a positive culture in the last 3 months.

Clinically stable with no significant changes in health status within 14 days prior to Screening or Day 1 Subjects are willing and able to perform requirements of the study.

Exclusion Criteria:

Smoking history in the prior 6 months Significant hemoptysis within 30 days prior to screening (>5 ml of blood in one coughing episode or >30 ml of blood in a 24 hour period) Forced expiratory volume at one second (FEV1) <40% of predicted On supplemental oxygen or SaO2 <90% at screening or Day 1, or within 30 days prior to enrollment.

Known cardiac (left heart) insufficiency (defined as LVEF <35%) prior to screening Known pulmonary hypertension Known or suspected hemoglobinopathy Initiation of NTM treatment regimen or a change in the regimen was made in the prior 6 months. Subjects on active treatment can be enrolled if they have been on a stable anti-NTM regimen for at least 6 months.

Initiation of new chronic therapy within 4 weeks prior to screening Use of drugs known to increase methemoglobin (see 12.2.7) at screening

Any of the following abnormal lab values at screening:

6-GPD deficiency Hemoglobin <10g/dl Platelet count <100,000/mm3 Prothrombin time international ratio (INR) >1.5 Abnormal liver function defined as any two of the following ALT >3x ULN AST >3x ULN ALP >3x ULN GGT >3x ULN

Abnormal renal function defined as:

Calculated Creatinine Clearance <50 ml (as calculated by Cockcroft/Gault)

For women of child bearing potential:

Positive pregnancy test at screening or Lactating or Unwilling to practice a medically acceptable form of contraception from screening to Day 15 (acceptable forms of contraception: abstinence, hormonal birth control, intrauterine device, or barrier method plus a spermicidal agent) Use of an investigational drug within 30 days prior to screening Intravenous or oral steroids (>10 mg/d prednisone equivalent) in the 14 days prior to screening Any condition that the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the subject.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Flume, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Oregon Health and Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Nitric Oxide (gNO): Participants will be treated for 3 weeks (5 days per week), Monday through Friday, and followed monthly for 3 months.
  The treatment period includes a physical exam, vital signs, blood tests, echocardiogram, spirometry test, sputum sample, questionnaires, and the inhalation gas treatment. During the inhalation gas treatment, participants will wear a face mask (similar to an oxygen mask) and will be given nitric oxide gas through the participants nose for three treatments with fifty minutes each time. They will then be followed up monthly during the Follow-up period with tests that include a physical exam and questionnaires.
Period: Overall Study
Arm/Group | Inhaled Nitric Oxide (gNO)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Inhaled Nitric Oxide (gNO)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.7 (24.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Patients With Negative Sputum Culture
Description: Sputum culture will be assessed for any sputum growth. A negative culture represents no mycobacterial growth.
Time Frame: End of Treatment (Day 15)
Measure: Number; unit: percentage of participants
Arm/Group | Inhaled Nitric Oxide (gNO)
Number analyzed (Participants) | 10
percentage of participants | 40
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide (gNO); This was a single arm trial. there is no comparator group; Test type: Other — Since no hypothesis testing was planned, no power analysis was required; Non Applicable; Non Applicable; The overall response rates were calculated, and exact binomial confidence intervals was constructed

2. Secondary Outcome: Number of Participants With Treatment Related Adverse Events as Assessed by the CTCAE (Common Terminology Criteria for Adverse Events)
Description: Adverse Events will be assessed by patient reporting and routine lab work
Time Frame: Treatment Day 1 through End of Treatment (3 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | Inhaled Nitric Oxide (gNO)
Number analyzed (Participants) | 10
Participants | 6

3. Secondary Outcome: Number of Participants With a Reduction in Semiquantitative Cultures
Description: Semiquantitative Culture Score is an assessment of bacterial burden with a lower score suggesting a lesser bacterial burden. The Semiquantitative Culture Score at Day 15 was compared to baseline, and a reduction in the Semiquantitative Culture Score suggests a reduced bacterial burden with treatment.
  Cultures were reported as positive if growth occurs in broth medium only; growth on broth medium plus solid medium cultures with countable colonies will be reported as 0-49 colonies, 1+; solid medium growth with 50-99 colonies, 2+; solid medium growth with 100-199 colonies; 3+, solid medium growth with 200-299 colonies; and 4+, solid medium growth with at least 300 colonies. For data analysis, each culture was scored as follows: 0, no growth in broth or solid medium; 1, broth medium growth only; 2, countable colonies (<50 colonies) on solid medium; and 3-6, 1+ to 4+ growth on solid medium, respectively.
Time Frame: At day 15 from baseline
Measure: Number; unit: participants
Arm/Group | Inhaled Nitric Oxide (gNO)
Number analyzed (Participants) | 10
participants | 4
Statistical Analysis 1: Comparison: Inhaled Nitric Oxide (gNO); This was a single arm trial. there is no comparator group; Test type: Other — Since no hypothesis testing was planned, no power analysis was required; The overall response rates were calculated, and exact binomial confidence intervals was constructed

ADVERSE EVENTS:
Time Frame: Patients were assessed for AE's throughout the duration of the study, approximately 3 months
Groups:
- Inhaled Nitric Oxide (gNO): evaluate the efficacy and safety of open-label exposure of gNO in patients with NTM lung disease
  gNO: This is a proof-of-concept study in which all subjects will be treated with gNO (i.e. no control) to see if there can be a microbiological effect by conversion to negative sputum cultures and how long that effect can be sustained following treatment.
Arm/Group | Inhaled Nitric Oxide (gNO)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (gNO) (N=10)
Transient Ischemic Attack (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhaled Nitric Oxide (gNO) (N=10)
Chest tightness (Cardiac disorders) | 1 (2)
Cough increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hematochezia (Gastrointestinal disorders) | 1 (2)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Nausea (Gastrointestinal disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Pain/pleurisy (Nervous system disorders) | 2 (2)
Shingles (Infections and infestations) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03748992/Prot_SAP_000.pdf